CLINICAL TRIAL: NCT04255615
Title: The Use of Artificial Intelligence for Clinical Assessment of Assisted Reproductive Techniques and IVF Outcomes
Brief Title: Use of Artificial Intelligence for Clinical Assessment of Assisted Reproductive Techniques and IVF Outcomes
Acronym: AI in ART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-06020306
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Infertility; in Vitro Fertilization (IVF); ART
Keywords: Artificial Intelligence
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D Ultrasound with AI (Other): AI tool to assess antral follicle count using 3 D Ultrasound
  Interventions: Other: AI to analyze 3 D ultrasound

INTERVENTIONS:
Other: AI to analyze 3 D ultrasound — AI to assess 3 D ultrasound to assess antral follicle count
  Other Names: z

SUMMARY:
The use of machine learning techniques using an artificial intelligence tool is proposed to analyze clinical data to predict best possible IVF/ART outcomes. This tool has been utilized to accurately predict embryo quality here at Cornell. Utilizing this tool to assess objective clinical findings and predict outcomes of assisted reproductive techniques is sought, with the ultimate goal of an automated tool to reduce implicit physician bias. Within this goal, using this tool to objectively and accurately assess baseline ovarian reserve at the start of an ART cycle is proposed, using 3D sonography to image the ovary and artificial intelligence tool to objectively identify baseline antral follicle counts.

DETAILED DESCRIPTION:
This study will collect prospective data, specifically 3D transvaginal ultrasound of ovaries at time of baseline evaluation at beginning of an ART cycle. All participants will be asked to give written consent to be included in the study. At the time of initial ultrasound that is routinely done on the first day of the ART cycle, the physician performing the ultrasound will use a 3D ultrasound transvaginal probe to perform the ultrasound and capture both 2D and 3D images. 3D ultrasound is performed routinely for patients undergoing ART and is not an investigative procedure, however is not uniformly performed at the time of the baseline ultrasound. As per standard practice, the baseline antral follicle count will be documented by the performing physician, as well as a 3D image saved to be analyzed later using AI.

Information about the medical history, treatment and outcomes will be collected as part of the study. Data maintained in the medical record as a result of standard of care monitoring for IVF and IUI will also be used for this study. This will include semen analysis (male partners if applicable) and pregnancy outcomes. For male partners, the semen analysis record will be part of the fertility history and semen analysis will be performed as standard of care with semen processing for fertilization. Additional data related to the treatment and outcomes will be collected from the medical record from the time of consent through the end of the treatment (including pregnancy outcomes).

The time commitment for subjects may take up to 1 month (time from consent signing to 3D ultrasound) and to the time of delivery if pregnant (up to 9 months). No further procedures will be performed in the study group.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing ovarian stimulation (including OI and IVF cycles)
* Treatment for fresh embryo transfer and cryopreservation of oocytes or embryos upfront
* Healthy male partners of the female subjects who agree to be part of the study.

Exclusion Criteria:

* None

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females undergoing IVF and their partners
Enrollment: 4000 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of baseline antral follicle count | Baseline
  To assess the accuracy and feasibility of using our artificial intelligence tool to assess antral follicle count, an indicator of baseline ovarian reserve, at time of baseline ultrasound for ART compared to qAVCantral and manual follicle counts to number of total oocytes retrieved.
Number of retrieved oocytes | 2 weeks
  To assess the accuracy and feasibility of using our artificial intelligence tool

SECONDARY OUTCOMES:
Number of mature oocytes | 2 weeks
  Number of mature oocytes (ART cycles)
Number of multiple gestation | approximately 6- 8 weeks
  Number of multiple gestation for OI cycles.
Number of clinical intrauterine pregnancies IVF | approximately 6- 8 weeks
  Clinical intrauterine pregnancies
Number of clinical intrauterine pregnancies OI | Approximately 6- 8 weeks
  Clinical intrauterine pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Nikica Zaninovic, PHD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No